CLINICAL TRIAL: NCT03927924
Title: Evaluation of the Effectiveness of High-intensity Focused Ultrasound for the Treatment of Prostate Cancer
Brief Title: High-intensity Focused Ultrasound Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: due to funding
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chi Hang Yee, Honorary Associate Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRE 2018.556
Record Dates: First submitted 2019-04-22; First posted 2019-04-25 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-06

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Focal Therapy; High-intensity focused ultrasound
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- High-intensity focused ultrasound (Experimental)
  Interventions: Procedure: High-intensity focused ultrasound

INTERVENTIONS:
Procedure: High-intensity focused ultrasound — Energy employed to exert its effect through thermal and mechanical destruction of cancer tissue

SUMMARY:
Conventional treatment options for localized prostate cancer include prostatectomy, radiotherapy and active surveillance. However, prostatectomy and radiotherapy carry certain degree of morbidity, including the risks of urinary incontinence, erectile dysfunction and injury to the structures in the proximity. Active surveillance carries the risk of disease progression and psychological distress to the patients. Focal therapy employs the concept of only destroying the significant lesion, resulting in disease cure and improved functional outcome. Among the different options of focal therapy, high-intensity focused ultrasound (HIFU) is one of the most commonly employed energy sources. It exerts its effect through thermal and mechanical destruction of cancer tissue. This study aims at assess the effectiveness of such treatment in prostate cancer management.

In this study, investigators evaluate the early oncological outcome and objective functional outcome of patients undergoing HIFU for the treatment of localized intermediate risk prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Visible index lesion(s) on MRI
* Index lesion(s) greater than 0.5 cm3
* Found to have localized low-risk or intermediate-risk prostate cancer after MRI-USG fusion targeted biopsy and saturation biopsy:

  1. Clinical tumour stage T2, or
  2. Gleason score 7, or
  3. PSA 20 ng/ml

Exclusion Criteria:

* Prostate size larger than 50 ml
* Patients unfit for contrast MRI exam
* Patients with previous treatment of prostate cancer
* Patients with previous surgery on the prostate
* Patients with active urinary tract infection
* Patients with bladder pathology including bladder stone and bladder cancer
* Patients with urethral stricture
* Patients with neurogenic bladder and/or sphincter abnormalities
* Fail to give informed consent

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only man will develop prostate cancer
Enrollment: 5 (Actual)
Dates: Start 2019-06-25 (Actual); Primary Completion 2021-01-28 (Actual); Study Completion 2021-01-28 (Actual)

PRIMARY OUTCOMES:
Absence of Prostate Cancer on Biopsy | 3 months
  Oncological outcome 1: percentage in absence of prostate cancer on biopsy

SECONDARY OUTCOMES:
Change in Urodynamic | 3 months and 6 months
  Functional outcome 1: change in urodynamic function assessed by flowrate
Change in Urinating Symptom Score | 3 months and 6 months
  Functional outcome 2: change in total scores in International Prostate Symptom Score (IPSS) questionnaires
Presence of Significant Prostate Cancer | 3 months
  Oncological outcome 2: presence of significant prostate cancer, defined by presence of Gleason score (ranges from 6 to 10) equals or more than 7
Change in Prostate specific antigen (PSA) | 3 months and 6 months
  Oncological outcome 3: PSA change after treatment
Pain score | Post treatment (day 1)
  Post-treatment pain score ranges from 1 to 10
Change in Prostate Symptom Score | 3 months and 6 months
  Functional outcome 3: change in symptom scores in EPIC-26 questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No